CLINICAL TRIAL: NCT02676986
Title: Phase II Window of Opportunity Study of Short-term Preoperative Treatment With Enzalutamide (Alone or in Combination With Exemestane) in Patients With Primary Breast Cancer
Brief Title: Short-term Preoperative Treatment With Enzalutamide, Alone or in Combination With Exemestane in Primary Breast Cancer
Acronym: ARB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 009684QM; 2014-002001-37 (EudraCT Number)
Record Dates: First submitted 2016-02-01; First posted 2016-02-09 (Estimated); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Primary Breast Cancer ER+ve; Primary Breast Cancer AR+ve TNBN
Keywords: Primary Breast Cancer; ER; AR; TNBC
MeSH Terms: interventions — enzalutamide; exemestane

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort I (ER positive cohort) (Active Comparator): Approximately 180 patients with ER positive breast cancer will be randomised 2:1 in favour of enzalutamide to receive enzalutamide plus exemestane or exemestane alone.
  Interventions: Drug: Enzalutamide; Drug: Exemestane
- Cohort II (AR positive, TNBC cohort) (Active Comparator): 55 patients with AR positive, TNBC will receive single agent treatment with enzalutamide.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — Anti-androgen
Drug: Exemestane — Hormonal therapy (Licenced)
  Arms: Cohort I (ER positive cohort)

SUMMARY:
Open-label, international, multicentre window of opportunity phase II trial to evaluate the effects of short-term preoperative therapy with enzalutamide (alone or in combination with exemestane) in women with newly diagnosed invasive primary breast cancer. The study has two cohorts:

* ER+ve breast cancer
* AR+ve, Triple-negative (i.e. ER-negative, PR-negative and HER2-negative) breast cancer

Study treatment is planned for a minimum of 15 days and a maximum of 29 days unless there is evidence of unacceptable toxicity or the patient requests to be withdrawn from the trial. Thereafter, patients will either be considered for definitive surgery or primary medical treatment (e.g. neoadjuvant chemotherapy) at the discretion of the treating physician.

The effects of enzalutamide (alone or in combination with exemestane) will be assessed on tumour tissue specimens taken at baseline and on the last day of study treatment.

ELIGIBILITY:
Main Inclusion Criteria:

1. Written informed consent prior to admission to this study
2. Female, aged ≥18 years
3. ECOG performance status 0- 2
4. Histologically confirmed invasive primary breast cancer
5. Palpable breast tumour of any size, or tumour with an ultrasound or MRI size of at least 1.0 cm
6. Haematologic and biochemical indices within the ranges shown below at the screening visit

   1. ANC 1500 cells/μl
   2. Platelet count 100000/μl
   3. Serum creatinine concentration < 1.5 x ULN
   4. Bilirubin level < 1.5 x ULN
   5. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) <3 x ULN

Inclusion Criteria unique to the ER+ve cohort:

1. ER+ve tumours defined as ≥1% of tumour cells positive for ER on IHC staining or an IHC score (Allred) of ≥3
2. Postmenopausal defined as:

   1. Age 55 years and 1 year or more of amenorrhea
   2. Age 55 years and 1 year or more of amenorrhea with LH and/or FSH levels in the postmenopausal range
   3. Age 55 with prior hysterectomy but intact ovaries with LH and/or FSH levels in the postmenopausal range
   4. Status after bilateral oophorectomy ( 28 days prior to first study treatment)

Inclusion Criteria unique to the AR+ve, TNBC cohort:

1. AR positive tumours defined as any nuclear AR staining by IHC (enrolment may be based on local pathology findings; subsequent review of AR expression by central pathology laboratory will be carried out)
2. Triple-negative tumours, i.e. tumour cells are negative for

   1. ER with <1% of cells positive on IHC or an IHC score (Allred) of ≤2
   2. PR with <1% of tumour cells positive on IHC or an Allred score of ≤2
   3. HER2 with 0, 1+ or 2+ intensity on IHC and no evidence of amplification of the HER2 gene on ISH
3. Negative serum or urine pregnancy test for women of childbearing potential within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible. Patients of childbearing potential must agree to use adequate contraception (for example, intrauterine device [IUD], birth control pills unless clinically contraindicated, or barrier device) beginning 2 weeks before the first dose of investigational medicinal product (IMP) and for 30 days after the final dose of IMP.

Exclusion Criteria:

1. Inflammatory breast cancer
2. Treatment with any of the following medications within 4 weeks before the baseline diagnostic biopsy is taken:

   1. Oestrogens, including hormone replacement therapy;
   2. Androgens (testosterone, dihydroepiandrosterone, etc.);
   3. Any approved or investigational agent that blocks androgen synthesis or targets the AR (e.g., abiraterone acetate, ARN-509, bicalutamide, enzalutamide, ODM-201, TAK-448, TAK-683, TAK-700)
3. Previous systemic or local treatment for the new primary breast cancer currently under investigation (including surgery, radiotherapy, cytotoxic and endocrine treatments); prior treatment for previous breast cancer or other neoplasms is allowed as long as it was completed at least 1 year prior to inclusion into this trial.
4. History of seizure or any condition that may predispose to seizure; history of loss of consciousness or transient ischemic attack within 12 months before day 1.
5. Significant cardiovascular disease, such as

   1. History of myocardial infarction, acute coronary syndromes or coronary angioplasty/stenting/bypass grafting within the past 6 months.
   2. Congestive heart failure New York Heart Association (NYHA) Class III or IV or history of congestive heart failure NYHA class III or IV, unless an echocardiogram or multigated acquisition scan performed within 3 months before day 1 reveals a left ventricular ejection fraction ≥ 45%;
   3. History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsade de pointes);
6. Hypersensitivity to the active pharmaceutical ingredient or any of the excipients of the IMPs, including Labrasol, butylated hydroxyanisole, and butylated Hydroxytoluene
7. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an IMP, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent.
8. Psychological, familial, sociological or geographical conditions that do not permit compliance with the study protocol.
9. Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational drug within 4 weeks prior to study entry.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2015-08-10 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Determine the difference in geometric mean change in Ki67 expression between the two treatment groups of patients in the ER+ Cohort | 24 months
  The geometric mean change will be determined by the change in Ki67 expression in tumour biopsy samples collected at the End of Treatment to those collected at Pre-Treatment
Determine the individual anti-proliferative response (RRΔKi67) for patients in the AR+ TNBC cohort | 24 months
  The anti-proliferative response is defined as a ≥50% fall in Ki67 expression over the course of the study treatment

SECONDARY OUTCOMES:
Determine the geometric mean change in Ki67 expression at the end of study treatment (Mean ΔKi67) for patients in the AR+ TNBC cohort | 24 months
Determine the geometric mean Ki67 expression at the end of study treatment (Mean Ki67post) for patients in the ER+ cohort | 24 months
Determine the individual end-of treatment anti-proliferative response (RRKi67-Post) for all patients. | 24 months
  The RRKi67-Post is defined as the natural logarithm of percentage positive Ki67 of less than 1 at the end of study treatment. For patients in the TNBC cohort, the analysis will be limited to patients with pre-treatment Ln (%Ki67) ≥ 1.
Determine the individual anti-proliferative response (RRΔKi67) for patients in the ER+ cohort. | 24 months
  The RRΔKi67 is defined as a ≥50% fall in Ki67 expression over the course of the study treatment
Determine the geometric mean change in Caspase-3 between end of study treatment and pre-treatment tumour samples (Mean ΔCaspase-3). | 24 months
Determine the individual apoptotic response (RRΔCaspase-3). | 24 months
  RRΔCaspase-3 is defined as a ≥50% increase in Caspase-3 over the course of the study treatment
Establish the safety and tolerability of enzalutamide alone and in combination with exemestane in this population through review of all AEs and SAEs assessed by CTCAE v4.03 | 24 months
  Safety and tolerability will be assessed through reviewing:
  * Incidence of serious adverse events (SAEs)
  * Incidence of grade 3 and 4 adverse events (AEs) (CTCAE, version 4.03)
  * Incidence of all AEs of all grades
  * Clinically significant changes in vital signs and clinical laboratory results during and following study drug administration
Measure the plasma levels of circulating hormones in blood samples collected prior to and at the end of study treatment. | 24 months
  Plasma levels of androstenedione, DHT, estradiol, estrone, estrone sulfate, follicle stimulating hormone, luteinizing hormone, progesterone, sex hormone binding globulin, and total/free testosterone will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schmid, Principal Investigator — Queen Mary University of London
Locations (41):
- MD Anderson Cancer Centre, Houston, Texas, United States
- Germany (28):
  - Evangelisches Krankenhaus Bergisch Gladbachg GmbH Frauenklinik, Bergisch Gladbach
  - Charité Campus Mitte, Berlin
  - Brustzentrum City St. Gertraudenkrankenhaus, Berlin
  - Evangelisches Waldkrankenhaus Spandau, Berlin
  - Johanniter Krankenhaus Bonn, Bonn
  - Onkologische Schwerpunktpraxis Bremen, Bremen
  - Klinikum Chemnitz GmbH, Chemnitz
  - Brustzentrum Uniklinik Köln, Cologne
  - St. Elisabeth Krankenhaus Köln, Cologne
  - Brustzentrum Holweide, Cologne
  - Kliniken-Essen-Mitte, Senology, Essen
  - Agaplesion Markus Krankenhaus, Frankfurt
  - Evangelische Kliniken Gelsenkirchen, Gelsenkirchen
  - Hannover Diakovere Henriettenstift, Hannover
  - Klinikum Kassel, Kassel
  - Klinikum Kempten, Kempten
  - UKSH -Campus Kiel, Kiel
  - DRK Kliniken Berlin Köpenick, Köpenick
  - UKSH Lübeck, Lübeck
  - UKSH Lüneburg, Städtisches Krankenhaus, Lüneburg
  - Johannes wesling Klinikum (Minden Hospital), Minden
  - Brustzentrum Niederrhein / ÜBAG Prof. Nitz Mönchengladbach, Mönchengladbach
  - Onkologisches Zentrum am Rotkreuzklinikum München, München
  - Helios-Kliniken Schwerin, Schwerin
  - Johanniter Frauenklinik Stendal, Stendal
  - Praxisnetzwerk Trosidorf, Troisdorf
  - GRN Klinik Weinheim, Weinheim
  - Marienhospital Witten, Witten
- Belfast Health and Social Care Trust, Belfast, Ireland
- Vall Hebron Hospital, Barcelona, Spain
- United Kingdom (10):
  - Royal Cornwall Hospitals NHS Trust, Truro, Cornwall
  - Ninewells Hospital and Medical School NHS Tayside, Dundee
  - Royal Devon and Exeter NHS Foundation Trust, Exeter
  - Barts Health NHS Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - University Hospital of South Manchester, Manchester
  - North Manchester Hospital, Pennine Acute Hospitals NHS Trust, Manchester
  - Churchill Hospital Oxford University Hospitals NHS Trust, Oxford
  - University Hospital of North Tees, Stockton-on-Tees
  - Royal Surrey County Hospital NHS Foundation Trust, Surrey

REFERENCES:
- See also: Clinical Study Report — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2014-002001-37